CLINICAL TRIAL: NCT02497521
Title: The German ADPKD Tolvaptan Treatment Registry is a Prospective, Observational, Multicentric Study of Patients Suffering From ADPKD That Are Considered for Tolvaptan Treatment.
Brief Title: The German ADPKD Tolvaptan Treatment Registry
Acronym: AD(H)PKD
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Roman Müller, MD, Prof., University Hospital of Cologne
Other Study IDs: 003
Record Dates: First submitted 2015-06-19; First posted 2015-07-14 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: ADPKD (Autosomal Dominant Polycystic Kidney Disease)
Keywords: polycystic kidney disease; autosomal dominant polycystic kidney disease; ADPKD; Tolvaptan; Jinarc
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADPKD: Patients with diagnosis of ADPKD, who are either evaluated for tolvaptan treatment indication, planned for tolvaptan treatment, or are already treated with tolvaptan

SUMMARY:
The German ADPKD Tolvaptan Treatment Registry is a prospective, observational, multicentric study of patients suffering from ADPKD that are considered for tolvaptan treatment. All ADPKD patients that are evaluated for treatment indication, or that are planned to be treated with tolvaptan, or that are already treated with tolvaptan are eligible. This registry is designed to provide "real-world" data on treatment management of patients with ADPKD.

DETAILED DESCRIPTION:
A substantial number of ADPKD patients treated in our center or referred to our center for counseling are considered eligible for tolvaptan treatment and, thus, will be invited to enter the registry. Furthermore, many patients with ADPKD are treated by nephrologists in practices. We operate a network with many of these practices and will expand this network. Patients can be enrolled - after having obtained approval by the local ethics committee - at external sites (expected number: about 500 patients per year). We are also closely liaised with the German self-help group PKDCure (PKD Familiaere Zystennieren e.V.), which is dedicated to ADPKD-linked research. Recruitment of patients will be facilitated by intensified interacting with these groups. Usually, patients that are referred to our institution for evaluation or counseling are regularly seen once a year. No additional trial-related visits in our institution will be required which is in line with the observational nature of the trial. However, data recording is not restricted to parameters assessed at our center but does include also parameters assessed by the treating physician.

SOPs (Standard Operating Procedures) that include further diagnostic tests like MRI are applied routinely in ADPKD patient management in our institution. The data obtained from these tests will be entered in the registry.

At enrolment, clinical, laboratory data and imaging study findings are collected after obtaining informed consent. The parameters listed below constitute the core data set, additional parameters can be included if considered essential.

Clinical data:

* demographic data (sex, age, height, weight)
* family history
* genotype (if available)
* extrarenal ADPKD manifestations
* co-morbidities
* medication
* physical examination
* blood pressure
* no. of extrarenal and renal complications in the past 12 months (urinary tract infections, pain episodes, macrohematuria, kidney stones, hospital admissions, ...)

Laboratory parameters include primarily (but not exclusively):

* serum sodium
* serum potassium
* serum osmolality
* serum creatinine
* estimated glomerular filtration rate (eGFR)
* serum urea
* serum uric acid
* whole blood count
* liver enzymes, bilirubin
* urinary sodium (spot and 24h-urine)
* urinary potassium
* urinary osmolality
* urinary creatinine
* urinary urea
* urinary uric acid
* urinary protein

Imaging study parameters:

* MRI - TKV (Total Kidney Volume)
* ultrasound
* (CT-scan if available)

Registered patients will be provided with diaries for documentation of tolvaptan dose, adverse side effects etc. These diaries are collected on a yearly basis and the data are included in the registry. Additionally the patients will be asked to fill in a questionnaire regarding the current medication, complications of ADPKD etc. once a year as well as a commercially available SF-12 (quality of life assessment) form.

Data capture will be done at yearly intervals starting at 12 months after enrolment. It includes the biochemical parameters and imaging study findings that have been obtained over the precedent 12 months.

The following additional data will be obtained:

* prescribed tolvaptan dose within the precedent 12 months
* maximum dose of tolvaptan given in the precedent 12 months
* weight, blood pressure
* urine output
* adverse effects
* hospital admissions
* occurrence of kidney pain, haematuria, or urinary tract infection
* complications associated with extrarenal manifestations of ADPKD
* data from diaries and questionnaires as mentioned above

According to the observational character of this study, no additional blood samples, examinations or imaging studies are required per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ADPKD proven by positive family history and evidence of renal cysts or diagnosed by treating physician
* Presentation at our center for tolvaptan treatment indication, or tolvaptan treatment planned, or tolvaptan already started

Exclusion Criteria:

* Patients not capable of giving informed consent
* End stage renal disease requiring renal replacement therapy
* Patients receiving tolvaptan as "off-label use"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of ADPKD and therapy with tolvaptan
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Drug dosing and titration as a measure of changes in real-life setting | 10 years
  Drug dosing and titration as a measure of maximum dose and the final dose and how fast it is achieved
Urine osmolarity as a measure of appropriate dosing | 10 years
  Data on urine osmolarity will be collected to measure appropriate dosing to provide the desired protective effect
Evaluation of rate of drug discontinuation and average Duration of therapy | 10 years
  Evaluation of rate of drug discontinuation and average Duration of therapy

SECONDARY OUTCOMES:
Demographics | 10 years
  Data on demographics will be collected
Clinical and biochemical characteristics at enrolment and treatment initiation | 10 years
Clinical and biochemical characteristics during follow-up | 10 years
Urinary output | 10 years
Evolution of estimated glomerular Filtration rate (eGFR) over the Observation period | 10 years
Evolution of TKV | 10 years
Side effects | 10 years
Liver enzymes | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Benzing, MD, Prof., Principal Investigator — University Hospital of Cologne; Roman-Ulrich Müller, MD, Prof., Principal Investigator — University Hospital Cologne
Locations (12):
- Germany (12):
  - Fachinternistische Gemeinschaftspraxis Markgraeferland, Müllheim, Baden-Wurttemberg
  - University Hospital of Wuerzburg, ZIM, Würzburg, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Nieren- und Diabeteszentrum Nettetal-Lobberich, Nettetal, North Rhine-Westphalia
  - University Hospital of Leipzig, Nephrologische Ambulanz, Leipzig, Saxony
  - Praxisgemeinschaft Dr. Peschel, Leipzig, Saxony
  - University Hospital of Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Nierenzentrum Lübeck, Lübeck, Schleswig-Holstein
  - University Hospital of Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Robert-Bosch-Krankenhaus, Stuttgart

REFERENCES:
- [Derived] Woestmann F, Strubl S, Farowski F, Arjune S, Tsakmaklis A, Todorova P, Spath MR, Brodesser S, Baar T, Grundmann F, Vehreschild MJGT, Muller RU. The Gut Microbiome in Autosomal Dominant Polycystic Kidney Disease: A Cross-Sectional Study. Kidney360. 2025 Nov 1;6(11):1906-1917. doi: 10.34067/KID.0000000836. Epub 2025 Jun 3. PMID 40459942
- [Derived] Bais T, Knol MGE, Xue L, Geertsema P, Vart P, Reichel F, Arjune S, Muller RU, Dekker SEI, Salih M, Meijer E, Gansevoort RT; DIPAK Consortium. Predicting Kidney Outcomes in Autosomal Dominant Polycystic Kidney Disease: A Comprehensive Biomarker Analysis. Clin J Am Soc Nephrol. 2025 May 1;20(5):608-618. doi: 10.2215/CJN.0000000680. Epub 2025 Mar 11. PMID 40067938
- [Derived] Arjune S, Lettenmeier K, Todorova P, Spath MR, Majjouti M, Mahabir E, Grundmann F, Muller RU. Inflammatory Cytokine Levels in Patients with Autosomal Dominant Polycystic Kidney Disease. Kidney360. 2024 Sep 1;5(9):1289-1298. doi: 10.34067/KID.0000000000000525. Epub 2024 Jul 24. PMID 39046800
- [Derived] van Heugten MH, Blijdorp CJ, Arjune S, van Willigenburg H, Bezstarosti K, Demmers JAA, Musterd-Bhaggoe U, Meijer E, Gansevoort RT, Zietse R, Hayat S, Kramann R, Muller RU, Salih M, Hoorn EJ; DIPAK Consortium. Matrix Metalloproteinase-7 in Urinary Extracellular Vesicles Identifies Rapid Disease Progression in Autosomal Dominant Polycystic Kidney Disease. J Am Soc Nephrol. 2024 Mar 1;35(3):321-334. doi: 10.1681/ASN.0000000000000277. Epub 2023 Dec 11. PMID 38073039
- [Derived] Woznicki P, Siedek F, van Gastel MDA, Dos Santos DP, Arjune S, Karner LA, Meyer F, Caldeira LL, Persigehl T, Gansevoort RT, Grundmann F, Baessler B, Muller RU. Automated Kidney and Liver Segmentation in MR Images in Patients with Autosomal Dominant Polycystic Kidney Disease: A Multicenter Study. Kidney360. 2022 Dec 29;3(12):2048-2058. doi: 10.34067/KID.0003192022. eCollection 2022 Dec 29. PMID 36591351
- See also: Portal for patients and referring physicians — https://www.adpkd.org/